CLINICAL TRIAL: NCT00318890
Title: A Phase I/II Trial of Induction Cisplatin and Docetaxel Followed by Concomitant Docetaxel/Radiotherapy With Subcutaneous Amifostine for Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: Cisplatin and Docetaxel Plus Docetaxel and Radiotherapy With Amifostine for Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Lisle Nabell, Primary Investigator, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F020522012; UAB 0210 (Other: Institutional study protocol number)
Record Dates: First submitted 2006-04-25; First posted 2006-04-27 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Cancer of Head and Neck; Head Cancer; Head and Neck Cancer; Neck Cancer; Neck Neoplasms
Keywords: Chemotherapy and Radiotherapy for Head and Neck Cancer; Chemotherapy, Radiotherapy Squamous Cell Carcinoma Head Neck
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cisplatin; Docetaxel; Radiotherapy; Amifostine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel + cisplatin followed by radiation (Experimental): Docetaxel with cisplatin is given for three cycles, followed by concomitant therapy with weekly docetaxel for 4 weeks. Radiation therapy is given 5 days each week on Days 64-106 with a concomitant boost in the last 2 weeks of treatment. Amifostine is given as an injection on a daily basis during radiotherapy.
  Interventions: Drug: Cisplatin; Drug: Docetaxel; Procedure: Radiotherapy; Drug: Amifostine

INTERVENTIONS:
Drug: Cisplatin — Cisplatin is given at a dose of 75 mg/m2 intravenously for three cycles on Days 1, 21, and 43.
  Other Names: Platinol-AQ
Drug: Docetaxel — Docetaxel is given at a dose of 75 mg/m2 intravenously on Days 1, 21, and 43 and continued at variable doses for 4 weeks with standard radiotherapy.
  Other Names: Taxotere
Procedure: Radiotherapy — Radiation therapy will be given 5 days each week for 4 weeks plus a concomitant boost in the last 2 weeks of treatment to deliver 54 Gy in 30 fractions. Radiotherapy will follow the induction chemotherapy with docetaxel and cisplatin.
Drug: Amifostine — Amifostine will be administered as a subcutaneous injection on a daily basis during radiotherapy.
  Other Names: Ethyol

SUMMARY:
This trial seeks to accomplish both local and regional control of head and neck cancer and reduce systemic metastatic disease. To do this, patients will received chemotherapy followed by chemotherapy and radiation (given together) with an escalating dose of docetaxel.

DETAILED DESCRIPTION:
The majority of head and neck cancer patients present with more advanced stages III or IV disease. The treatment of cancers of the head and neck can have profound consequences with regard to functional abilities such as speech and eating. In the treatment of both locally advanced HNSCC and sites where organ preservation is desirable, radiation therapy has been a major method of treatment. However, as a single modality, radiation therapy can cure fewer than 30% of patients with advanced disease. Attempts to improve the outcome of locally advanced HNSCC have generally added chemotherapy to radiotherapy. However, the optimal manner to integrate chemotherapy into the plan of care has been controversial. Chemotherapy has been used most commonly as either induction therapy preceding radiation, or more recently as concomitant therapy along with radiation. Induction chemotherapy has been associated with high response rates of 60-90%, but no significant change in loco-regional control or survival.Clinical trials incorporating chemotherapy with concurrent radiation have recently generated considerable interest. To accomplish both loco-regional control and reduce systemic metastasis, this trial proposes induction chemotherapy followed by concomitant chemotherapy-radiation with an escalating dose of docetaxel in patients with locally advanced previously untreated HNSCC.

ELIGIBILITY:
Inclusion Criteria:

* The patient has histologically proven primary or recurrent squamous cell carcinoma arising in the oropharynx, oral cavity, hypopharynx, larynx, or nasopharynx.
* The patient has stage III or IV disease.
* Performance status < 2 (ECOG scale) with a life expectancy of > 12 months.
* Age 19 years and above.
* The patient is medically fit to tolerate a course of definitive radiation therapy.
* The patient has:

  1. adequate hepatic function with bilirubin < upper limit of normal (ULN)
  2. transaminases (SGOT and SGPT) may be up to 2.5 x ULN if alkaline phosphatase is < ULN, or alkaline phosphatase may be up to 4 x ULN if transaminases are < ULN
  3. adequate renal function with serum creatinine < 1.5 mg/dl (or estimated creatinine clearance of > 50 mL/min)
  4. normal serum calcium
  5. adequate hematologic function as: defined by an absolute neutrophil count > 1500/ml, hemoglobin > 8.0 g/dl, and platelet count > 100,000/ml.
* The patient may have had a prior malignancy but must be three years from treatment.
* A history of superficial non-melanoma skin cancer or in situ carcinoma of the cervix less then three years will be allowed.
* The patient must agree to use effective contraception if procreative potential exists, and continue contraception for at least 6 months following completion of the study.
* Patient must sign informed consent.

Exclusion Criteria:

* The patient has received radiation therapy previously to the head and neck.
* The patient has received prior chemotherapy for head and neck cancer.
* The patient is pregnant or lactating.
* Peripheral neuropathy > Grade 2.
* Serious non-malignant disease (e.g. congestive heart failure, uncontrolled atrial fibrillation, active hepatitis).
* Any underlying psychological condition that would prohibit the understanding and rendering of informed consent.
* Patients with a history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80 must be excluded.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2002-10; Primary Completion 2007-04 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To establish the response rate to chemotherapy followed by docetaxel with radiotherapy and to assess overall survival, local-regional recurrence rate and effects on the quality of life. | approximately 4 months

SECONDARY OUTCOMES:
To evaluate the toxicities of chemotherapy followed by concomitant docetaxel with radiotherapy in patients. | approximately 4 months
To evaluate tumor specimens for intermediary biomarkers of response or prognosis as compared to normal tissue | approximately 4 months
To assess the tolerance to subcutaneous amifostine and its effect on saliva production. | approximately 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Lisle Nabell, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States